CLINICAL TRIAL: NCT02136498
Title: Internet-based Medication Adherence Program for Nicotine Dependence Treatment
Brief Title: My Mobile Advice Program: A Randomized Pilot Feasibility Study
Acronym: MyMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Michigan (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34DA034612 (NIH)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Smoking Cessation; Medication Adherence
Keywords: smoking cessation; varenicline; adherence
MeSH Terms: conditions — Smoking Cessation; Medication Adherence | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mHealth self-help + varenicline (Active Comparator): Participants in this control arm received standard cognitive-behavioral self-help materials delivered via a mobile health (mHealth) program + a standard course of varenicline.
  Interventions: Drug: Varenicline; Behavioral: Cognitive-behavioral self-help
- mHealth MyMAP program + varenicline (Experimental): Participants in the experimental arm received standard cognitive-behavioral self-help materials delivered via a mHealth program + additional personalized support features (automated, tailored advice managing nicotine withdrawal symptoms and medication side-effects & secure messaging with a cessation counselor; i.e., MyMAP program) + a standard course of varenicline.
  Interventions: Drug: Varenicline; Behavioral: Cognitive-behavioral self-help; Behavioral: MyMAP (My Mobile Advice Program)

INTERVENTIONS:
Drug: Varenicline — Standard 12 week course of varenicline, provided in both arms
  Other Names: Chantix
Behavioral: Cognitive-behavioral self-help — Standard self-help education for smoking cessation, delivered via mobile-optimized website accessible via smartphone.
Behavioral: MyMAP (My Mobile Advice Program) — Same standard self-help intervention as in control arm + automatically-tailored support and advice for managing nicotine withdrawal symptoms + secure messaging with cessation counselor
  Arms: mHealth MyMAP program + varenicline

SUMMARY:
The purpose of this pilot study is to evaluate the acceptability and feasibility of the proposed smoking cessation intervention (called MyMAP or My Mobile Advice Program).

DETAILED DESCRIPTION:
Investigators will develop and pilot test a prototype of the MyMAP intervention.The intervention is designed to help smokers better manage issues known to reduce treatment adherence (withdrawal symptoms, medication side-effects, low motivation, and inadequate behavioral skills for medication adherence) and to facilitate greater communication between patients and providers so clinicians can provide appropriate oversight of medication use, intervene when medically necessary, and address patient concerns that may otherwise lead to non-adherence or early treatment termination.

ELIGIBILITY:
Inclusion Criteria:

* An invited member of Group Health, a health care system in the Pacific Northwest
* Plan to remain enrolled in Group Health for the next 6 months
* aged 18 - 65
* Eligible for smoking cessation treatment through Group Health insurance coverage
* smoke >= 10 cigs a day
* speak and read in English
* willing to use varenicline and no contraindications for this medication
* ready to quit smoking
* have a smart phone with internet access
* willing to receive study texts and emails
* receive care at a Group Health clinic and have electronic medical records in this system
* fill prescriptions through the Group Health pharmacy
* agree to use birth control while taking study medication, if there is a risk of pregnancy

Exclusion Criteria:

* lifetime history of dementia
* psychosis or bipolar disorder based on self-report or medical record review
* hearing, comprehension or visual limitations that preclude full study participation
* current use of other forms of tobacco
* any medical contraindication for varenicline use
* documented history of suicidal ideation/intent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McClure, PhD, Principal Investigator — Group Health Research Institute; Sheryl Catz, PhD, Principal Investigator — University of California, Davis; Larry An, MD, Principal Investigator — University of Michigan
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McClure JB, Anderson ML, Bradley K, An LC, Catz SL. Evaluating an Adaptive and Interactive mHealth Smoking Cessation and Medication Adherence Program: A Randomized Pilot Feasibility Study. JMIR Mhealth Uhealth. 2016 Aug 3;4(3):e94. doi: 10.2196/mhealth.6002. PMID 27489247
- See also: Primary outcome paper — http://dx.doi.org/10.2196/mhealth.6002

RESULTS

PARTICIPANT FLOW:
Groups:
- mHealth Self-help + Varenicline: Participants in the control arm received standard self-help education delivered via an mHealth program (accessible via smart phone) and a prescription for a standard 12 week course of varenicline.
  Standard self-help included topics such as: how to make a quit plan, how to use varenicline, how to manage cravings to smoke, how tot manage nicotine withdrawal and medication side-effects, relapse prevention, etc.
- mHealth MyMAP + Varenicline: Participants in the experimental arm received a mHealth program (accessible via smartphone) and a prescription for a standard 12 week course of varenicline.
  The mHealth intervention included the same self-help content offered to controls + a) real-time, adaptively-tailored advice for managing nicotine withdrawal symptoms and medication side-effects and b) asynchronous secure messaging with a cessation counselor.
Period: Overall Study
Arm/Group | mHealth Self-help + Varenicline | mHealth MyMAP + Varenicline
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mHealth Self-help + Varenicline | mHealth MyMAP + Varenicline | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (8.9) | 48.4 (8.4) | 49.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31 | 30 | 61
  Non-white | 2 | 3 | 5
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes] | 16.9 (4.5) | 18.5 (9.1) | 17.7 (7.2)
Prior use of varenicline [Number; unit: participants]
  Used varenicline previously | 14 | 14 | 28
  Never used varenicline | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence Abstinence
Description: Self-report of no-smoking, even a puff during the last 7 days.
Time Frame: 5 month follow-up
Population: Intent to treat analyses with missing cases imputed as smokers.
Measure: Number; unit: Percentage of people not smoking
Groups:
- Augmented mHealth Self-help + Varenicline: Participants in the experimental arm received a mHealth program (accessible via smartphone) and a prescription for a standard 12 week course of varenicline.
  The mHealth intervention included the same self-help content offered to controls + a) real-time, adaptively-tailored advice for managing nicotine withdrawal symptoms and medication side-effects and b) asynchronous secure messaging with a cessation counselor.
Arm/Group | mHealth Self-help + Varenicline | Augmented mHealth Self-help + Varenicline
Number analyzed (Participants) | 33 | 33
Percentage of people not smoking | 24 | 36

2. Secondary Outcome: Number of Days of Varenicline Use
Description: Number of days varenicline was used
Time Frame: 5 mo follow-up
Measure: Mean (Standard Deviation); unit: Mean number of days
Arm/Group | mHealth Self-help + Varenicline | Augmented mHealth Self-help + Varenicline
Number analyzed (Participants) | 33 | 33
Mean number of days | 39 (28.9) | 46 (31.9)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study period (~ 6 months).
Description: Medication side-effects/nicotine withdrawal symptoms (adverse events) were assessed at each follow-up using a standard checklist of events, resulting in a high number of reports in both arms. Experimental participants were also asked to report ongoing side-effects and symptoms to receive tailored treatment advice, increasing reports in this arm.
Arm/Group | mHealth Self-help + Varenicline | mHealth MyMAP + Varenicline
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/33
Other Adverse Events (participants affected / at risk) | 30/33 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mHealth Self-help + Varenicline (N=33) | mHealth MyMAP + Varenicline (N=33)
Passive suicidal ideation without intent (Psychiatric disorders) | 0 (0) | 1 (1) — Participant reported passive suicidal ideation (without intent) on his wedding anniversary from his estranged wife. Participant had a history of psychiatric issues and was not taking varenicline at the time.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mHealth Self-help + Varenicline (N=33) | mHealth MyMAP + Varenicline (N=33)
Anger or irritability (Psychiatric disorders) | 11 (12) | 15 (24)
Anxiety (Psychiatric disorders) | 8 (9) | 8 (12)
Change in appetite (Gastrointestinal disorders) | 15 (23) | 9 (16)
Confusion/difficulty concentrating (Psychiatric disorders) | 6 (7) | 8 (12)
Constipation (Gastrointestinal disorders) | 5 (6) | 5 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 13 (16)
Craving to smoke (Psychiatric disorders) | 22 (40) | 30 (74)
Depression (Psychiatric disorders) | 2 (2) | 4 (7)
Diarhhea (Gastrointestinal disorders) | 5 (6) | 3 (4)
vivid or unusual dreams (General disorders) | 21 (24) | 19 (36)
Drowsiness (General disorders) | 4 (4) | 2 (2)
Gas (Gastrointestinal disorders) | 13 (14) | 15 (33)
Headache (General disorders) | 11 (12) | 12 (23)
Insomnia or trouble sleeping (General disorders) | 12 (13) | 18 (33)
Nausea (Gastrointestinal disorders) | 10 (11) | 11 (15)
Rapid heart beat or chest pain (General disorders) | 0 (0) | 2 (3)
stomach pain or vomiting (Gastrointestinal disorders) | 9 (10) | 7 (8)
Memory problems (Psychiatric disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
The primary limitation of this pilot study is the small sample size, which prevents definitive conclusions about the efficacy of the MyMAP intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No